CLINICAL TRIAL: NCT01932892
Title: Quantifying Prosthetic Socket Interface Movement
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 20130075
Record Dates: First submitted 2013-05-08; First posted 2013-08-30 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Transhumeral Amputation
Keywords: transhumeral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transhumeral prosthesis user: Transhumeral body-powered prosthesis user

SUMMARY:
This study will quantify motion occurring at the socket interface of transhumeral prosthesis users during common tasks. Participants in the study will use a body powered prosthesis with a hosmer hook terminal device. A motion analysis system and a novel optical sensor embedded into the socket wall will record the amount of movement between the residual limb and socket of the prosthesis. Participants will complete range of motion and functional tasks. The range of motion tasks include shoulder flexion, abduction and rotation as well as elbow flexion. The functional tasks include bilateral lift of weighted basket, unilateral lift of weighted handle, box and blocks test, walk and carry a gallon of milk, and folding a towel. It is expected that the more weight at the terminal device the more rotation at the interface, as well as more slip between residual limb and device. It is also expected that the soft tissues of the residual limb can be modeled as a nonlinear spring and the amount of movement at the interface can be predicted based off the force in the system.

DETAILED DESCRIPTION:
Participation in the study will begin at the socket duplication stage/initial testing phase and end no more than a week later after the second collection day is complete. Subjects will meet individually with the PI at lab on testing day one to have their socket duplicated and do some initial testing. Socket duplication will consist of filling the inside volume of the socket with a plaster mixture to form a positive mold. Once set, this positive mold can be removed and used by a contractor to form the clear thermoplastic socket over it. After the mold has been made, the subject will perform a series of tasks while being recorded by an 8 camera Vicon motion analysis system and 2 digital video cameras. Thirty reflective markers will be placed on the subject using an adhesive collar. There is slight risk of skin irritation due to the adhesive tape, similar to wearing a Band-Aid. Some discomfort may arise while removing the markers. A tight fitting shirt will be worn by participants to limit undesired motion of the markers due to loose clothing. Subjects will complete:

* Range of Motion Trials (without prosthesis)

  o The Range of Motion (ROM) trials include shoulder flexion/extension, shoulder abduction/adduction, and shoulder rotation. Each RoM task will be repeated three times.
* Trinity Amputation and Prosthesis Experience Scales (TAPES)
* This questionnaire looks at different aspects of having and using a prosthesis.
* Results of this questionnaire will be compared to performance in the laboratory setting to see the correlation between how the user rates the device and how the perform with it.

The first collection day will last about 1-2 hours. For the second collection day, subjects will be randomized into group A or B to determine the order of sockets tested during data collection on the second day. Subjects in group A will use their original prosthesis in the first collection while group B subjects will use their duplicate socket prosthesis. Subjects will switch to the other socket for the second collection session. The second day is expected to last about 3-4 hours. Each session will consist of the following:

* Range of Motion Trials (with prosthesis)

  o The RoM trials include shoulder flexion/extension, shoulder abduction/adduction, shoulder rotation, and elbow flexion/extension. Each RoM task will be repeated three times.
* Functional Tasks
* Unilateral lift

  * Subject will pick and place a series of weights from one spot on a 3' high shelf to another spot 3' away on the same shelf. The participant must hold the object above the shelf (cannot drag the object) during the transfer and the weight of the object will be varied from 5 to 25lbs in 5lbs increments.
  * Amount of movement at the socket interface and time to complete each transfer will be evaluated using this task. We expect that more socket interface movement will
* Bilateral lift

  * Subject will lift a basket containing a series of weights from the floor to a 3' high shelf, and then back to the original position. The weight in the basket will be varied from 10 to 50lbs in 10lbs increments.
  * Maximum load transferred, and time to complete each transfer will be evaluated using this task. We expect time to complete task will translate to ability to appropriately position the devise. Weight lifted serve as a strength control for the unilateral lift.
* Walk and Carry

  * Participants will walk on a treadmill for 1 minute while carrying a 15 pound bag.
  * The amount of slip and socket rotation will be recorded.
* Cut play-dough with knife and fork

  * Participants sit in front of a table with a plate of play-dough. Participants will be allowed to pick up and use the knife and fork however they desire, but must cut the play dough into three roughly even pieces. This task will be repeated 3 times.
  * The time to complete the task, and which hand is used to hold the knife, will be used to determine capability for dexterous manipulation.
* Folding a towel

  * Participants will stand before a bath towel laid flat on a table. Subjects will fold the towel in half lengthwise, then in half widthwise, then in half lengthwise. This task will be repeated 3 times.
  * The time to complete the task will be used to determine capability for dexterous manipulation.
* Modified Box and Blocks Test

  * 16 blocks will be placed in 4 rows on one side of a box with a partition in the middle. The objective is to move one block at a time to the other side going over the partition. Participants will be instructed to start at the lower right corner and complete that row before moving to the next. Subjects will move each block to the matching spot on the opposite half of the box. Participants will have 1 minute to move as many blocks as they can. Participants will repeat this task 4 times. The box will start placed so the blocks start on the same side as the participants prosthesis.
  * Outcomes from this test will include the number of blocks moved in the allotted time or the time required to move all 16 blocks, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Transhumeral amputee
* Uses prosthesis
* Used same socket without documented skin condition for at least 2 months

Exclusion Criteria:

* Current skin condition on part of residual limb

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Magnitude of prosthetic socket rotation and slip | 3 hours
  Motion capture data and optical sensor data will be used to calculate the amount of prosthetic socket rotation and slip. It is predicted that current socket designs will have some degree of socket movement during normal activities due to soft tissue deformation.

SECONDARY OUTCOMES:
Magnitude of prosthetic socket movement relative to end effector loading | 3 hours
  Motion capture data and optical sensor data will be used to calculate the amount of socket movement compared to the terminal device loading for the various tasks. It is predicted that tasks which have more load at the terminal device will result in more socket movement.
Magnitude of prosthetic socket movement relative to the amount of residual limb rotation. | 3 hours
  The amount of socket movement will be compared to the amount of residual limb rotation for each task. Residual limb rotation is the angle between the upper arm segment and the scapula segment. It is hypothesized the greater the residual limb angle, the greater the amount of socket movement.
Difference in range of motion of the shoulder joint between no prosthesis, the original prosthetic socket, and the duplicate socket | 3 hours
  It is predicted that the range of motion of the shoulder will be statistically the same between the original and duplicate socket.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Carey, PhD, Study Director — University of South Florida
Locations (1):
- Rehabilitation Robotics and Prosthetics Testbed, Tampa, Florida, United States

REFERENCES:
- See also: Center for Assistive Rehabilitation Robotic Technologies — http://carrt.eng.usf.edu